CLINICAL TRIAL: NCT05629429
Title: Olaparib Maintenance Therapy in Patients With Metastatic Breast Cancer Following DNA-damaging Based Chemotherapy
Brief Title: Olaparib Maintenance Therapy in Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202202045MIPA
Record Dates: First submitted 2022-11-02; First posted 2022-11-29 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: olaparib treatment (Experimental): Olaparib 300mg BID PO
  Interventions: Drug: Olaparib
- Arm2: continuation of the chemotherapy (Active Comparator): continuation of the current platinum based chemotherapy
  Interventions: Drug: Chemotherapy drug

INTERVENTIONS:
Drug: Olaparib — Olaparib 300mg BID PO
  Arms: Arm 1: olaparib treatment
Drug: Chemotherapy drug — Continue platinum based chemotherapy
  Arms: Arm2: continuation of the chemotherapy

SUMMARY:
Olaparib, a PARP inhibitor, is proven as an effective therapy for germline BRCA1/2-mutated breast cancer; however, the therapeutic efficacy for somatic mutation in BRCA1/2 or genes of homologous recombination DNA repair is unclear. Maintenance of Oalaprib can delay the disease progression in patients with BRCA1/2 mutated advanced ovarian cancer after treatment with platinum based chemotherapy. The investigators design a phase 2 study to evaluate the efficacy of maintenance of Olaparib in patients with metastatic breast cancer. The investigators enroll patients with metastatic ER(+)Her2(-) or triple-negative breast cancer. Patients who are chemotherapy-naïve or prior 1-line chemotherapy are eligible for screening. All eligible patients will receive 4 cycles of platinum based chemotherapy. Gene test will be performed on their breast tumor. If patients have mutation of HR genes and at least stable disease after platinum based chemotherapy, they will be randomized to treatment arm (Olaparib maintenance) or control arm (continuation of chemotherapy). The primary end-point is progression-free survival, and the secondary end-point is to assess the response rate, overall survival and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a life expectancy ≥ 16 weeks.
2. Provision of informed consent prior to any study specific procedures
3. 20 years of age or older; gender includes female and male
4. ECOG 0-1
5. Patients should be diagnosed as metastatic breast cancer ER(+)Her2(-) or TNBC, diagnosis could be by local hospital
6. HER2 negative [IHC 0, 1+ or IHC 2+ with corresponding ISH non-amplified of ratio less than 2.0 or ISH nonamplified ratio less than 2.0] as per ASCO-CAP HER2 guideline recommendations 2013 (ASCO-CAP).
7. At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI)
8. Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1. Postmenopausal is defined at least one of the followings: (a) Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments; (b) Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post menopausal range for women under 50; (c) radiation- induced oophorectomy with last menses >1 year ago; (d) chemotherapy-induced menopause with >1 year interval since last menses; (f) surgical sterilisation (bilateral oophorectomy or hysterectomy)
9. Male patients must use a condom during treatment and for 3 months after the last dose of olaparib when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception ([see appendix H for acceptable methods]) if they are of childbearing potential
10. No more than previous 0-1 line of chemotherapy after metastasis confirmed
11. For ER(+) breast cancer, patients should fail at least 1-line of hormone therapy (either in adjuvant setting or in metastatic cancer) before entering this study
12. Patients should undergo 4-cycles of platinum-based chemotherapy and have a CR, PS or SD prior to randomisation.
13. At least one measurable lesion that can be accurately assessed at baseline by computed tomography (CT) (magnetic resonance imaging [MRI] where CT is contraindicated) and is suitable for repeated assessment as per RECIST 1.1.
14. Patients must have normal organ and bone marrow function measured within 28 days prior to randomisation as defined below:

    1. Haemoglobin (Hb) ≥10.0 g/dL
    2. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    3. Platelet count ≥100 x 109/L
    4. Total bilirubin ≤1.5 x institutional upper limit of normal (ULN) unless the patient has documented Gilbert's Syndrome
    5. Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be ≤ 5x ULN
    6. Patients must have creatinine clearance (CrCl) of ≥51 mL/min estimated or measured using standard methodology at the investigating centre (i.e. Cockcroft-

Gault, MDRD, CK-EPI, EDTA or 24 hr urine):

-

Exclusion Criteria:

-

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

1. Cytotoxic chemotherapy, hormonal or non hormonal targeted therapy within 21 days of Cycle 1 Day 1 is not permitted. Palliative radiotherapy must have been completed 21 or more days before Cycle 1 Day 1. The patient can receive a stable dose of bisphosphonates or denosumab for bone metastases, before and during the study as long as these were started at least 5 days prior to study treatment.
2. More than 2 prior lines of cytotoxic chemotherapy for metastatic disease.

   1. Prior treatments with hormonal therapy and non hormonal targeted therapy are allowed and not counted as a prior line of cytotoxic chemotherapy.
   2. For the purposes of this protocol, the combination of "an aromatase inhibitor and everolimus" or "a hormonal therapy and CDK4/6 inhibitor" is not considered cytotoxic chemotherapy.
   3. Treatment with biologics will not be considered as prior line of therapy.
   4. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment
3. Previous treatment with a PARP inhibitor (including olaparib)
4. The minimum washout period for immune checkpoint blockade therapy shall be 21 days.
5. Patients with MDS/AML or with features suggestive of MDS/AML.
6. Patients with second primary cancer, EXCEPTIONS: adequately treated non melanoma skin cancer, curatively treated in-situ cancer of the cervix, Ductal Carcinoma in Situ (DCIS), stage 1 grade 1 endometrial carcinoma, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years prior to study entry (including lymphomas [without bone marrow involvement]).
7. Mean resting corrected QTc interval using the Fridericia formula (QTcF) >470 msec/female patients and >450 msec for male patients (as calculated per institutional standards) obtained from 3 ECGs performed 2-5 minutes apart at study entry, or congenital long QT syndrome.
8. Any of the following cardiac diseases currently or within the last 6 months

   1. Unstable angina pectoris
   2. Congestive heart failure ≥ Class 2 as defined by the New York Heart Association
   3. Acute myocardial infarction
   4. Conduction abnormality not controlled with pacemaker or medication (patients with a conduction abnormality controlled with pacemaker or medication at the time of screening are eligible)
   5. Significant ventricular or supraventricular arrhythmias (patients with chronic rate- controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible)
9. Concomitant use of known strong cytochrome P (CYP) 3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg.

   ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting study treatment is 2 weeks.

   Patient has had prescription or non-prescription drugs or other products known to be sensitive CYP3A4 substrates or CYP3A4 substrates with a narrow therapeutic index, or to be moderate to strong inhibitors/inducers of CYP3A4 which cannot be discontinued 2 weeks prior to Day 1 of dosing and withheld throughout the study until 2 weeks after the last dose of study drug. Patients should stop using herbal medications 7 days prior to first dose of study treatment.
10. Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting study treatment is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
11. Persistent toxicities (≥ CTCAE grade 2) caused by previous cancer therapy, excluding alopecia.
12. Major surgery within 2 weeks of starting study treatment: patients must have recovered from any effects of any major surgery.
13. Immunocompromised patients, eg, patients who are known to be serologically positive for human immunodeficiency virus (HIV).
14. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection.

    a. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution CT scan or any psychiatric disorder that prohibits obtaining informed consent, and any other medical condition that, in the opinion of the Investigator, places the patient at unacceptable risk of toxicity.
15. Patients with symptomatic uncontrolled brain metastases.

    1. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease (SD) for 28 days.
    2. Patients with a history of treated central nervous system (CNS) metastases are eligible, provided they meet all of the following criteria: Disease outside the CNS is present. No clinical evidence of progression since completion of CNS-directed therapy. Minimum of 3 weeks between completion of radiotherapy and Cycle 1 Day 1 and recovery from significant (Grade ≥3) acute toxicity with no ongoing requirement for >10 mg of prednisone per day or an equivalent dose of other corticosteroid. If on corticosteroids, the patient should be receiving a stable dose of corticosteroids, started at least 4 weeks prior to treatment.
16. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
17. Patients with a known hypersensitivity to olaparib or any of the excipients of the products.
18. Pregnant or breast feeding women.
19. Patients with HBV infection and uncontrolled hepatitis are not eligible. If patients are HBV carriers (HBsAg-positive without 2.5x elevation of AST/ALT), these patients can enter study if they have baseline HBV-DNA level assessed during screening, receive prophylactic medication and regularly monitored by GI doctor. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
20. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
21. Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable, for timing refer to inclusion criteria no.7

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
CT or MRI assessment | 3 years
  Progression-free survival

SECONDARY OUTCOMES:
Survive or death | 3 years
  Overall survival rate
CT or MRI assessment | 3 years
  Response rate
Questionnaire | 3 years
  Quality of life

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - National Taiwan University Hospital, Taipei, Please Select
  - Taipei Veterans General Hospital, Taipei, Please Select
  - National Taiwan University Hospital Yunlin branch, Yuanlin